CLINICAL TRIAL: NCT02529930
Title: An Exploratory Safety and Immunogenicity Study of Human Papillomavirus (HPV16+) Immunotherapy VB10.16 in Women With High Grade Cervical Intraepithelial Neoplasia (HSIL; CIN 2/3)
Brief Title: An Exploratory Safety and Immunogenicity Study of HPV16+ Immunotherapy VB10.16 in Women With HSIL; CIN 2/3)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Theradex (Industry); Vaccibody AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VB C-01
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: High Grade Cervical Intraepithelial Neoplasia
Keywords: HSIL; CIN 2/3; Therapeutic DNA vaccine; Human Papillomavirus; Immunotherapy
MeSH Terms: interventions — Vaccines, DNA; Biological Products; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: 3mg VB10.16 Vaccine (Experimental): VB10.16 Immunotherapy (DNA vaccine): Biological/Vaccine Vaccination time points: Week 0, Week 3, Week 6, 3mgs per vaccination
  Interventions: Biological: VB10.16 Immunotherapy (DNA vaccine)
- Cohort 2: 3mg VB10.16 Vaccine (Experimental): VB10.16 Immunotherapy (DNA vaccine): Biological/Vaccine Vaccination time points: Week 0, Week 4, Week 8, 3mgs per vaccination
  Interventions: Biological: VB10.16 Immunotherapy (DNA vaccine)

INTERVENTIONS:
Biological: VB10.16 Immunotherapy (DNA vaccine) — Patients will receive 3 vaccinations of 3 mg VB10.16 at the pre-specified time points. VB10.16 will be administered intramuscularly in the area over the lateral deltoid muscle.
  Other Names: Biological/Vaccine

SUMMARY:
This is an exploratory, open, prospective multi-centre study of VB10.16 immunotherapy in patients with high grade HPV16+ Cervical Intraepithelial Neoplasia (HSIL; CIN2/3). This study will recruit approximately 27-40 female patients with high grade cervical intraepithelial neoplasia (HSIL, CIN 2/3) at multiple sites in Europe.

DETAILED DESCRIPTION:
The study will be divided into two phases, a dosing and expansion phase.

During the dosing phase the safety, tolerability and immunogenicity of 2 different vaccination schedules of 3 mg VB10.16 immunotherapy will be established in a minimum of 12 patients with histology confirmed CIN 2.

During the expansion phase the safety, tolerability and immunogenicity of the selected vaccination schedule will be evaluated in approximately 15 to 20 patients with histology confirmed HPV16+ CIN 2/3.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Women ≥18 years
2. Women with ectocervical HPV16+ associated High Grade Cervical Intraepithelial Neoplasia (HSIL) as verified by local pathology:

   (Dosing Phase: Women with histologically confirmed HPV16+ associated CIN 2; Expansion Phase: Women with histologically confirmed HPV16+ associated CIN 2/3)
3. Satisfactory colposcopic examination.

Exclusion Criteria (abbreviated):

1. More than 2 cervical quadrants of CIN 3 as visualised by colposcopy.
2. Atypical glandular cells (AGC) or adenocarcinoma in situ (AIS) on cytology, malignant cells on cytology or histology or other suspicion of either micro-invasive or invasive disease.
3. Current severe pelvic inflammatory disease, severe cervicitis, or other severe gynaecological infection as per colposcopy and clinical examination.
4. Positive serological test for hepatitis C virus or hepatitis B virus surface antigen (HBsAg) or human immunodeficiency virus (HIV).
5. Administration of any blood product within 3 months of enrolment.
6. Concomitant or prior malignant disease.
7. Clinically significant autoimmune disease.
8. Known allergy to Kanamycin or other aminoglycosides
9. Known immunodeficiency and or immunosuppression.
10. History of toxic shock syndrome.
11. Evidence or history of clinically significant cardiac disease
12. Active infection requiring parenteral antibiotics.
13. Tattoos, scars, or active lesions/rashes within 2 cm of the site of vaccination or any implantable leads.
14. Immunosuppression
15. Major surgery within 3 months of trial entry.
16. Current or recent (within 30 days of first study treatment) participation in a clinical trial.
17. Previous vaccination (either therapeutic and/or prophylactic) against HPV.
18. Administration of any live vaccine within 90 days of trial entry.
19. Concomitant anticancer therapies.
20. Inadequate bone marrow function
21. Inadequate liver function
22. Clinical significant electrolyte abnormalities
23. Women of childbearing age not willing to use an effective form of contraception
24. Pregnancy or intention to become pregnant
25. Nursing women
26. Evidence of any other medical condition that may interfere with study participation, patient compliance or place the patient at high risk from treatment-related complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability | 6 months (extended follow up for additional 6 months)
  - The percentage of patients with adverse events (AEs), including any dose-limiting toxicities (DLT), laboratory assessments and physical findings.

SECONDARY OUTCOMES:
Immunogenicity | 6 months
  * The percentage of patients with E6/E7 specific cellular immune response in the blood.
  * The percentage of patients with cellular immune response in the target lesions.
  * The percentage of patients with humoral response against the E6/E7 viral antigen.
Preliminary assessment of efficacy | 6 months (extended follow up for additional 6 months)
  * The percentage of patients with HPV16+ clearance.
  * The percentage of patients with lesion regression

CONTACTS AND LOCATIONS:
Overall Officials: Irene Skjørestad, MSc, Study Director — Vaccibody AS
Locations (4):
- Germany (4):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Lower Saxony
  - IZD Institut für Zytologie und Dysplasie, Hanover, Lower Saxony
  - Medical School Hanover, Hanover, Lower Saxony
  - Klinikum Wolfsburg, Wolfsburg, Lower Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillemanns P, Denecke A, Woelber L, Bohmer G, Jentschke M, Schjetne KW, Bruins Slot KMH, Fredriksen AB. A Therapeutic Antigen-Presenting Cell-Targeting DNA Vaccine VB10.16 in HPV16-Positive High-Grade Cervical Intraepithelial Neoplasia: Results from a Phase I/IIa Trial. Clin Cancer Res. 2022 Nov 14;28(22):4885-4892. doi: 10.1158/1078-0432.CCR-22-1927. PMID 36129459